CLINICAL TRIAL: NCT01002274
Title: Open-Label, 40-weeks Extension of Protocol MCS-2-TWN-a to Further Evaluate the Efficacy and Safety of MCS-2 for the Treatment of Lower Urinary Tract Symptoms Suggestive of Benign Prostatic Hyperplasia in Treatment Naïve Male Subjects
Brief Title: Open-Label Extension Study of MCS-2 in the Treatment of Lower Urinary Tract Symptoms
Acronym: MCS-2-TWN-c
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCS-2-TWN-c
Record Dates: First submitted 2009-10-21; First posted 2009-10-27 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; BPH; MCS-2; Multi-Carotenoids; Lower Urinary Tract Symptoms; International prostate symptom score
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCS-2 (Experimental): 2 soft-gel capsules Qd for 40 weeks
  Interventions: Drug: MCS-2

INTERVENTIONS:
Drug: MCS-2 — 2 soft-gel capsules Qd for 40 weeks
  Other Names: MUS

SUMMARY:
This is an open-label extension study of another study protocol, MCS-2-TWN-a. Subjects who have completed the 12-week treatment and procedures under the protocol MCS-2-TWN-a will be eligible for this study.

DETAILED DESCRIPTION:
This open-label extension study is designed to further assess the long-term safety and efficacy of MCS-2. Subjects who have completed the 12-week treatment and procedures under the protocol MCS-2-TWN-a will be eligible for another 40 weeks of MCS-2 treatment at the same daily dosage as the active treatment given under the protocol MCS-2-TWN-a. Subjects are limited to those who are currently not being treated medically for BPH or LUTS.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed 12 weeks of treatment under the protocol MCS-2-TWN-a.
* Subject is able to understand and willing to conform to the study procedures and has signed the informed consent form for participation in this extension study.

Exclusion Criteria:

* Subject has severe LUTS at the last visit under the protocol MCS-2-TWN-a.
* Subject is considered ineligible for the study by the investigator(s).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 40 weeks

SECONDARY OUTCOMES:
Changes from baseline in International Prostate Symptom Scores (I-PSS) | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan